CLINICAL TRIAL: NCT03159208
Title: Prediction of Functional Outcomes From Chronic Critical Illness
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Duke University (Other); University of Pittsburgh (Other); University of Washington (Other); University of Colorado, Denver (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0998; R01NR016459 (NIH)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Chronic Critical Illness; Prolonged Mechanical Ventilation
Keywords: Prognosis; Critical Illness; Ventilation, Mechanical; Disease Attributes; Socioeconomic Factors; Activities of Daily LIving; Cognition
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration; Disease Attributes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to establish clinical determinants of poor cognitive and physical functional outcome of CCI patients so that the investigators may develop and validate a multi-dimensional clinical prediction model to more effectively inform decision making earlier in the course of the ICU care. The investigators hypothesize that multiple premorbid and acute factors measured early in the course of CCI will have strong independent associations with functional recovery. The investigators further hypothesize that social and economic factors are associated with long-term functional outcomes independent of the acute clinical problems.

DETAILED DESCRIPTION:
A substantial number of critically ill patients experience persistent organ failure leading to chronic critical illness (CCI). The majority of these patients die within a year, and many survivors must cope with long-term physical and cognitive limitations that are often severe. Survival with severe physical and cognitive dysfunction is a significant clinical, emotional, and economic burden in this population, but little is known about which patients are at highest risk for physical and cognitive dysfunction. Moreover, although long-term mortality in CCI can be reliably estimated with a validated mortality prediction model, there is currently no validated method to predict long-term functional disability for purposes of shared decision-making and resource planning. In order to address these gaps in knowledge, the investigators will conduct a multi-center prospective cohort study that measures clinical and premorbid risk factors for long-term physical and cognitive dysfunction in CCI. Using these risk factors, the investigators will construct a multi-outcome prognostic model for survival with severe physical or cognitive dysfunction to facilitate shared decision-making and resource planning. Additionally, the investigators will identify independent social and economic variables that are risk factors for long-term survival and functional disability.

ELIGIBILITY:
Inclusion Criteria

1. Patients in enrolling ICU
2. Expected to require 7 days of mechanical ventilation uninterrupted for 72 hours for acute illness.
3. Adults >/= 18yo of age.

Exclusion Criteria

1. Patients with respiratory failure due to neuromuscular disease
2. Patients with respiratory failure due to severe burn
3. Patients requiring chronic mechanical ventilation at home
4. Patients receiving mechanical ventilation at an outside hospital >7 days
5. Expected death prior to day 8 of mechanical ventilation therapies in 24 hrs.
6. Prisoners
7. No family member or surrogate available
8. Patient not proficient in English (or Spanish at select sites)
9. Unwilling or unable to provide written informed consent (patient or when indicated, by surrogate)
10. Co-enrollment in another study not approved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at risk for chronic critical illness after prolonged mechanical ventilation for acute illness or injury.
Sampling Method: Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients who Survive with Severe Physical Disability | 12 months
  Severe Physical Disability defined by requiring assistance with 4 of 6 or more Activities of Daily Living (ADLs).
Proportion of Patients who Survive with Severe Cognitive Disability | 12 months
  Severe Cognitive Disability defined by the Informant Questionnaire on Cognitive Delay (IQCODE) average score of greater than 3.44 (range 0-5, 5 being worse) and, when available, the Telephone Montreal Cognitive Assessment (T-MoCA) score of less than 17 (Range 0-22, 0 being worse). Severity of Cognitive Delay will be confirmed with a Functional Activities Questionnaire (FAQ) score of greater than 8 (Range 0-30, 30 being worst).
Proportion of Patients who Survive with Severe Physical and Cognitive Disability | 12 months
  Severe Physical Disability defined by requiring assistance with 4 of 6 or more Activities of Daily Living (ADLs). Severe Cognitive Disability defined by the Informant Questionnaire on Cognitive Delay (IQCODE) average score of greater than 3.44 (range 0-5, 5 being worse) and, when available, the Telephone Montreal Cognitive Assessment (T-MoCA) score of less than 17 (Range 0-22, 0 being worse). Severity of Cognitive Delay will be confirmed with a Functional Activities Questionnaire (FAQ) score of greater than 8 (Range 0-30, 30 being worst).
Proportion of Patients who Survive with No Severe Functional Disability | 12 months
  No severe physical disability is indicated by requiring assistance with 3 or fewer Activities of Daily Living (ADLs). No Severe Cognitive Disability is defined by the Informant Questionnaire on Cognitive Delay (IQCODE) average score of less than 3.44 (range 0-5) and, when available, the Telephone Montreal Cognitive Assessment (T-MoCA) score of greater than 17 (Range 0-22).
Proportion of patients who die within one year | 12 months
  Confirmed dead at 1-year follow up.

SECONDARY OUTCOMES:
Proportion of Patients who Survive with Severe Physical Disability | 6 months
  Severe Physical Disability defined by requiring assistance with 4 of 6 or more Activities of Daily Living (ADLs).
Proportion of Patients who Survive with Severe Cognitive Disability | 6 months
  Severe Cognitive Disability defined by the Informant Questionnaire on Cognitive Delay (IQCODE) average score of greater than 3.44 (range 0-5, 5 being worse) and, when available, the Telephone Montreal Cognitive Assessment (T-MoCA) score of less than 17 (Range 0-22, 0 being worse). Severity of Cognitive Delay will be confirmed with a Functional Activities Questionnaire (FAQ) score of greater than 8 (Range 0-30, 30 being worst).
Proportion of Patients who Survive with Severe Physical and Cognitive Disability | 6 months
  Severe Physical Disability defined by requiring assistance with 4 of 6 or more Activities of Daily Living (ADLs). Severe Cognitive Disability defined by the Informant Questionnaire on Cognitive Delay (IQCODE) average score of greater than 3.44 (range 0-5, 5 being worse) and, when available, the Telephone Montreal Cognitive Assessment (T-MoCA) score of less than 17 (Range 0-22, 0 being worse). Severity of Cognitive Delay will be confirmed with a Functional Activities Questionnaire (FAQ) score of greater than 8 (Range 0-30, 30 being worst).
Proportion of Patients who Survive with No Severe Functional Disability | 6 months
  No severe physical disability is indicated by requiring assistance with 3 or fewer Activities of Daily Living (ADLs). No Severe Cognitive Disability is defined by the Informant Questionnaire on Cognitive Delay (IQCODE) average score of less than 3.44 (range 0-5) and, when available, the Telephone Montreal Cognitive Assessment (T-MoCA) score of greater than 17 (Range 0-22).
Proportion of patients who die within 6 months. | 6 months
  Confirmed dead at 6 month follow up.
Patient Quality of Life Score: NeuroQOL | 6 and 12 months.
  Quality of Life with cognitive ability is measured by Quality of Life in Neurological Disorders (NeuroQOL) with 8-items Scores range from 8-20. The higher score indicates better health state perceived by participant.
Patient Quality of Life Score: EQ-5D | 6 and 12 months.
  Quality of Life is measured by EQ-5D Questionnaire via 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The score ranges from -0.594 to 1.000 in the US. The higher score indicates a better health state perceived by the participant.
Caregiver Quality of Life Score: EQ-5D | 6 and 12 months
  Quality of Life is measured by EQ-5D Questionnaire via 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The score ranges from -0.594 to 1.000 in the US. The higher score indicates a better health state perceived by the participant.
Caregiver Burden Score: BSFC | 6 and 12 months
  Caregiver burden is measured by the Burden Scale for Family Caregivers (BSFCs) with 10-items and are rated on a scale from 0 (strongly disagree) to 3 (strongly agree). The score ranges from 0 to 30 points. The higher scores indicate greater caregiver burden.
Caregiver Anxiety and Depression Score: HADS | 12 months
  Caregiver Depression and Anxiety is measured by the Hospital Anxiety and Depression Scale (HADS) with 14-items. Scores for each subscale (anxiety and depression) range from 0 to 21. Scores for the entire scale range from 0 to 42. The higher scores indicating more distress.
Caregiver PTSD Score: IES-R | 12 months
  Caregiver PTSD symptoms is measured by Impact of Events Scale-Revised (IES-R) with 22-items. Scores for each subscale (avoidance, intrusion, hyperarousal) range from 0-12. Scores for the entire scale range from 0-88. The higher scores are associated with clinical symptoms of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Carson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (6):
- United States (6):
  - Denver Health and Hospital Authority, Denver, Colorado
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset will be available to investigators 9-36 months following publication of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: Data can be obtained upon application to primary investigators. Investigators who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Hough CL, Caldwell ES, Cox CE, Douglas IS, Kahn JM, White DB, Seeley EJ, Bangdiwala SI, Rubenfeld GD, Angus DC, Carson SS; ProVent Investigators and the National Heart Lung and Blood Institute's Acute Respiratory Distress Syndrome Network. Development and Validation of a Mortality Prediction Model for Patients Receiving 14 Days of Mechanical Ventilation. Crit Care Med. 2015 Nov;43(11):2339-45. doi: 10.1097/CCM.0000000000001205. PMID 26247337
- [Background] Kahn JM, Le T, Angus DC, Cox CE, Hough CL, White DB, Yende S, Carson SS; ProVent Study Group Investigators. The epidemiology of chronic critical illness in the United States*. Crit Care Med. 2015 Feb;43(2):282-7. doi: 10.1097/CCM.0000000000000710. PMID 25377018
- [Background] Nelson JE, Cox CE, Hope AA, Carson SS. Chronic critical illness. Am J Respir Crit Care Med. 2010 Aug 15;182(4):446-54. doi: 10.1164/rccm.201002-0210CI. Epub 2010 May 6. PMID 20448093